CLINICAL TRIAL: NCT06990594
Title: A Multi-Center Bidirectional Cohort Study on Total Knee Arthroplasty for the Treatment of Knee Osteoarthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, YujiakuoTHU, Prof., Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 25034-0-02
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: A total of 120 participants will be enrolled, with 40 receiving total knee arthroplasty (TKA) using a personalized prosthesis, 40 receiving semi-personalized TKA, and 40 receiving conventional TKA. Participants will be followed for one year post-surgery to assess clinical outcomes.

SUMMARY:
The purpose of this study is to evaluate the clinical benefits of different types of total knee arthroplasty (TKA) in osteoarthritis treatment. The study aims to compare surgical outcomes, functional recovery, complication rates, and cost-effectiveness among personalized, semi-personalized, and conventional TKA in a multi-center, bidirectional cohort study.

DETAILED DESCRIPTION:
This study aims to assess the performance of personalized, semi-personalized, and conventional total knee arthroplasty (TKA) procedures across different patient groups.

This is a prospective cohort and controlled study involving 120 patients, including 40 in the experimental group receiving personalized TKA, 40 receiving semi-personalized TKA, and 40 in the control group receiving conventional TKA. Participants will be 50-80 years old, diagnosed with end-stage knee osteoarthritis, post-traumatic arthritis, avascular necrosis, inflammatory arthritis, or deformities requiring total knee arthroplasty. They will be followed for one year post-surgery to assess clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 50-80 years.
2. Diagnosed with end-stage knee osteoarthritis, post-traumatic arthritis, avascular necrosis, or inflammatory arthritis requiring total knee arthroplasty.
3. Willing and able to provide informed consent.

Exclusion Criteria:

1. History of prior knee surgery or knee replacement.
2. Severe knee deformity (valgus >20° or varus >15°) or instability.
3. Severe contracture (>25° flexion contracture).
4. Undergoing total knee revision surgery.
5. Rheumatoid arthritis diagnosis.
6. BMI >35.
7. Neuromuscular disorders affecting knee stability or gait.
8. Pregnancy or lactation.
9. Presence of significant comorbidities posing unacceptable risk.
10. Active or recent severe infections or malignancy.
11. History of drug or alcohol abuse in the past six months.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of 120 patients aged 50-80 years diagnosed with end-stage knee osteoarthritis, post-traumatic arthritis, avascular necrosis, or inflammatory arthritis, who require total knee arthroplasty (TKA). Participants will be recruited from multiple centers, including Beijing Tsinghua Chang Gung Hospital, Peking University Shougang Hospital, and Beijing Chaoyang Hospital. The study will compare personalized, semi-personalized, and conventional TKA procedures in terms of surgical outcomes, functional recovery, complication rates, and cost-effectiveness.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score (KSS) | At baseline, 6 months, and 12 months post-surgery
  The KSS is a standardized assessment tool used to evaluate knee function and pain following total knee arthroplasty. It includes an objective knee score and a functional score, measuring alignment, stability, and range of motion.

SECONDARY OUTCOMES:
Pain Severity | At baseline, 6 months, and 12 months post-surgery
  Visual Analog Scale (VAS) and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be used to assess pain levels pre- and post-surgery.
Functional Improvement | At baseline, 6 months, and 12 months post-surgery.
  Functional improvement will be measured using SF-36 Health Survey, Knee Injury and Osteoarthritis Outcome Score (KOOS), and gait analysis.
Prosthesis Positioning and Alignment | At baseline and 12 months post-surgery.
  Radiographic evaluation will assess implant positioning and limb alignment.
Surgical Complication Rate | At 12 months post-surgery.
  The rate of postoperative complications including infections, deep vein thrombosis (DVT), and revision surgeries will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China